CLINICAL TRIAL: NCT05246553
Title: Electrical Stimulation of the Peripheral Vestibular System in Order to Develop a Vestibular Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nils Guinand (Other)
Collaborators: University of Geneva, Switzerland (Other); Maastricht University Medical Center (Other); Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor-Investigator, Nils Guinand, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NAC 11-080 CER 11-129
Record Dates: First submitted 2022-01-14; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Vestibular Disorder; Bilateral Vestibulopathy; Bilateral Vestibular Loss
Keywords: Vestibular; Prosthesis; Otorhinolaryngologic Diseases; Electrical Stimulation; Vestibular Implant
MeSH Terms: conditions — Vestibular Diseases; Bilateral Vestibulopathy; Otorhinolaryngologic Diseases | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Modified cochlear implant recipients (Experimental): Patients suffering from severe to profound hearing loss and severe bilateral vestibulopathy implanted with a modified cochlear implant providing 1 to 3 extracochlear electrodes implanted in proximity to the ampullary branches of the vestibular nerve (vestibular electrodes).
  All experiments will be carried out while the vestibular electrodes are inactive, and while electrical stimulation is delivered to one or several vestibular electrodes, with and without concurrent cochlear stimulation.
  Interventions: Procedure: Electrical stimulation of the vestibular system; Procedure: Electrical stimulation of the auditory system
- Cochlear Implant Patients (CI) (Active Comparator): Unilateral or bilateral cochlear implant recipients with normal vestibular function documented within the clinical follow up of their cochlear implant, and without previous history of vestibular symptoms or complaints.
  Interventions: Procedure: Electrical stimulation of the auditory system
- Bilateral vestibulopathy Patients (BV) (Active Comparator): Patients with documented diagnosis of bilateral vestibulopathy, according to the guidelines of the Barany society (Strupp et al., Journal of Vestibular Research, vol. 27, no. 4, pp. 177-189, 2017).
  Interventions: Diagnostic Test: Bilateral vestibulopathy Patients (BV)
- Unilateral vestibulopathy Patients (UV) (Active Comparator): Patients with documented diagnosis of unrecovered unilateral vestibulopathy, consistent with the current classification of vestibular disorders of the Bárány Society (www.jvr-web.org/ICVD.html).
  Interventions: Diagnostic Test: Unilateral vestibulopathy Patients (UV)
- Healthy Subjects (HS) (No Intervention): Normal auditory functiona and without previous auditory or vestibular symptoms or complaints. Normal vestibular function documented with the video-head impulse test.

INTERVENTIONS:
Procedure: Electrical stimulation of the vestibular system — Patients are implanted with a modified cochlear implant (CI) which comprises one to three extracochlear electrodes that are placed in the proximity of vestibular afferents (i.e., vestibular nerves or the ampullae of each semicircular canal), and an intracochlear array. Trains of electrical stimulation in the form of charge-balanced, biphasic pulses can be delivered through each of the implanted electrodes (cochlear or vestibular) and modulated via computer-controlled signals, audio signals (captured with a microphone) or by signals captured by head-mounted motion sensors.
  Other Names: Vestibular implant
  Arms: Modified cochlear implant recipients
Procedure: Electrical stimulation of the auditory system — A cochlear implant (CI) is a device providing a sense of sound to a person who suffers from severe to profound sensorineural hearing loss. A CI comprises the following parts, a microphone (capturing the sound from the environment), a speech processor (receiving and encoding the sounds captured by the mircophone), a transmitter-receiver antenna pair (transmitting the information from the external to the implanted components), an implanted stimulator (converting the signal into a tonotopically arranged set of electrical pulses) and an electrode array inserted in the cochlea that will deliver the electrical pulses to different portions of the auditory nerve. Trains of electrical stimulation in the form of charge-balanced, biphasic pulses can be delivered through each of the electrodes in the cochlear array and modulated via computer-controlled signals or audio signals (captured with a microphone).
  Other Names: Cochlear implant
  Arms: Cochlear Implant Patients (CI); Modified cochlear implant recipients
Diagnostic Test: Bilateral vestibulopathy Patients (BV) — Diagnosis established on the basis of the consensus document of the Classification Committee of the Bárány Society (Strupp et al., Journal of Vestibular Research, vol. 27, no. 4, pp. 177-189, 2017).
  Arms: Bilateral vestibulopathy Patients (BV)
Diagnostic Test: Unilateral vestibulopathy Patients (UV) — Patients with documented diagnosis of unrecovered unilateral vestibulopathy, consistent with the current classification of vestibular disorders of the Bárány Society (www.jvr-web.org/ICVD.html).
  Arms: Unilateral vestibulopathy Patients (UV)

SUMMARY:
This study has three main goals (1) to explore the effects of electrical stimulations of the peripheral vestibular system(2) to assess the potential of this technique to rehabilitate basic vestibular functions in patients with severe bilateral vestibulopathy, and (3) to take advantage of the unprecedented experimental paradigm provided by the vestibular implant to increase our fundamental knowledge on the contribution of peripheral vestibular function to posture, gait and higher order sensory functions, mechanisms that remain poorly understood.

DETAILED DESCRIPTION:
The investigators will carry out a thorough investigation of the effects of electrical stimulation on vestibular and auditory function in a group of patients implanted with a modified cochlear implant providing extracochlear electrodes implanted in the vicinity of the of the ampullary nerve branches. These results will be compared to similar measurements carried out in a group of age and sex-matched healthy controls, in a group of patients with bilateral and unilateral vestibulopathy, and also in a group of patients implanted with a cochlear implant and normal vestibular function. The protocol comprises the following specific measurements:

1. Clinical evaluation of auditory function: pure-tone and speech audiometry.
2. Clinical evaluation of vestibular function: clinical evaluation of the vestibulo-ocular reflex (e.g., video-nystagmography, video-head impulse tests), and of the otolithic function (vestibular evoked myogenic potentials).
3. Dynamic visual acuity: loss of visual acuity while walking in a treadmill at controlled speed, compared to the static (standing in place) of the subject.
4. Auditory and vestibular brainstem evoked potentials.
5. Electroencephalography.
6. Temporal Binding Window: maximal time interval separating two different types of sensory stimuli (visual, auditory and vestibular) within which the subject still perceives them as simultaneous.
7. Psychophysical motion detection tests: motion perception thresholds measured in a platform allowing specific and smooth motion profiles in 3 linear and 3 angular dimensions.
8. Gait and posture: functional gait assessment, postural sway in conditions providing accurate or conflicting sensory (e.g., vestibular, visual, proprioceptive) information.
9. Spatial navigation in real and virtual reality environments (e.g. Morris water maze, standardized clinical environment).
10. Monitoring of the autonomous nervous system: standard, non-invasive clinical investigations of cardiovascular, ophthalmic, secretory, or metabolic functions (e.g., blood pressure, heart rate, pupillary reflex).

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a vestibular implant showing neither auditory function nor vestibular one.
* Control group of patients implanted with a cochlear implant and presenting a normal vestibular function.
* Control group of patients with bilateral vestibular loss.
* Control group of patients with unilateral vestibular loss and finally
* Control group of healthy subjects with normal auditory and vestibular functions.

All sujbects included in the study will be older than 18 years old.

Exclusion Criteria:

* Children
* Patients suffering from blindness,
* Patients suffering from major ophtalmologic damage
* Patients suffering from neurologic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Vestibular Ocular Reflex (VOR) amplitude | Immediately after the vestibular electrodes are activated
  The canal function of the vestibular system is evaluated based on the VOR measurement.The participant is sited and wearing goggles with movement sensors allowing to measure head movement and a camera to record eyes movements (lightweight infrared eye tracker with built in 6 degree of freedom inertial measurement unit i.e eyeseecam). A trained examiner generates randomized head pulses toward the left or the right while the participant has to stare at a target in front of him. The ratio between head and eyes velocity (amplitude or "gain") is then calculated.
Change in Vestibular Ocular Reflex (VOR) threshold | Immediately after the vestibular electrodes are activated
  The canal function of the vestibular system is evaluated based on the VOR measurement.The participant is sited and wearing goggles with movement sensors allowing to measure head movement and a camera to record eyes movements (lightweight infrared eye tracker with built in 6 degree of freedom inertial measurement unit i.e eyeseecam). An electrical stimulation is generated using the vestibular implant and the velocity threshold for VOR is then quantified.
Changes in pure tone audiometry measurements | Immediately after the cochlear and/or vestibular electrodes are activated
  Pure tone audiometry presents pure (one-frequency) tones to each ear and determines the threshold of hearing for the participant. This test is performed in a sounfproof cabin with the patient sited.
Changes in speech audiometry measurements | Immediately after the cochlear and/or vestibular electrodes are activated
  The participant is sited in a soundproof cabin while wearing headphones. The participant hears a recording of a list of common words spoken at different volumes and is asked to repeat those words.
Changes in logatomes test results | Immediately after the cochlear and/or vestibular electrodes are activated
  Logatomes are nonsense syllables used for analyzing the confusion of phonemes.The participant is sited in a soundproof cabin while wearing headphones. The participant hears a recording of a list of logatomes with a structure of consonant-vowel-consonant (c-v-c) and vowel-consonant-vowel (v-c-v) and is asked to repeat those logatomes.
Changes in the Temporal Binding Window (TBW) | Immediately after the cochlear and/or vestibular electrodes are activated
  Different combinaisons of auditory, visual and vestibular stimuli are used to determine the respective TBW. The participants are sited in a chair and presented with two different stimuli. They are then asked which stimulus comes first. In patients implanted with a VI, the investigators specifically stimulate the vestibular system and pair this stimulation to a visual or auditory one. The time interval between the two stimuli is progressively decreased until they are percieved as simultaneous. It is thus possible to calculate the TBW.
Changes in the Auditory and Vestibular evoked potentials (AEPs-VEPs) | Immediately after the cochlear and/or vestibular electrodes are activated
  The participant is sited with eyes open. Electrophysiological responses are recorded during the presentation of brief and controlled stimulus. In subjects with a vestibular implant the evoked potentials are recorded following an electrical vestibular stimulation. An electrical cochlear stimulation is used for subjects with a cochlear implant. In healthy controls a brief sound or bone vibration is used.
Changes in the cortical and subcortical activity | Immediately after the vestibular electrodes are activated
  Electroencephalography (EEG) is a brain exploratory method the investigators will use to estimate the latency of evoked cortical and subcortical potentials following a visual, auditory and vestibular stimulation. The electrical signals are recorded using electrodes placed on the participant scalp.
Changes in the Vestibular Evoked Myogenic Potentials (VEMPs) | Immediately after the vestibular electrodes are activated
  For cervical-VEMP recording, a very brief electrical stimulation of the vestibular system is applied. The participant lies on an examination table and is asked to lift his head and turn it toward the stimulation opposite side in order to contract the sternocleidomastoid muscle (SCM) whose myogenic activity is recorded using surface electrodes. The stimulus is the same for ocular-VEMP recording. The sited participant is asked to keep his gaze up and the ocular muscles myogenic activity is recorded.
Changes in motion perception | Immediately after the vestibular electrodes are activated
  The participant is sited in a chair anchored to a six degrees of freedom motion platform. Stimuli are different types of movements. The participant is asked to mention if he perceives a movement and if so to eventually give its direction. The statistical analyses of these answers allow to determine a perception threshold for each type of movement.
Changes in gait dynamics while walking at different speeds | Immediately after the vestibular electrodes are activated
  Participant is asked to walk six meters straightforward at: normal, slow, and fast auto-selected speeds as well as the fastest speed possible. Changes in three-dimensional kinematics during the different tasks will be assessed using a 12-camera optoelectronic motion capture system. Participants will be equipped with 35 reflective markers placed on specific anatomical landmarks according to the full-body. The test is performed twice per participant within a 1-week interval, to allow reliability (test-retest) analyses.
Changes in gait dynamics performing the Timed "Up & Go" | Immediately after the vestibular electrodes are activated
  Partipants are sited on a chair. At the "Go" of the examinor they are asked to stand up, walk for three meters, make a u-turn, come back and sit back on the chair. Changes in three-dimensional kinematics during the different tasks will be assessed using a 12-camera optoelectronic motion capture system. Participants will be equipped with 35 reflective markers placed on specific anatomical landmarks according to the full-body. The test is performed twice per participant within a 1-week interval, to allow reliability (test-retest) analyses.
Changes in Functional Gait Assessment (FGA) performances | Immediately after the vestibular electrodes are activated
  The FGA is used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. The FGA comprises ten tasks during which changes in three-dimensional kinematics will be assessed using a 12-camera optoelectronic motion capture system. Participants will be equipped with 35 reflective markers placed on specific anatomical landmarks according to the full-body.The test is performed twice per subject within a 1-week interval, to allow reliability (test-retest) analyses.
Postural changes (sway threshold and/or amplitudes) | Immediately after the vestibular electrodes are activated
  The investgators will use a modified SMART EquiTest to implement a custom protocol developed to identify potential biomarkers of vestibular deficiency using pseudorandom stimulus waveforms to perturb balance. The device delivers continuous surface or visual surround rotations that evoke antero-posterior body sway in participants. The test starts with a 4 min warm-up in order to familiarize the participant with the environment. Then participants undergo 4-min test in 3 conditions: (1) surface-tilt stimuli with eyes closed, (2) surface-tilt with eyes open and visual surround fixed, and (3) visual surround tilt with fixed surface with all using 2° peak-to-peak stimulus amplitudes. Participants are also be equipped with a 3-DOF Head Tracker (part of the EquiTest system) continuously recording head movements in the Yaw, Pitch, and Roll planes. Postural assessments areperformed twice per participants within a 1-week interval, to allow reliability (test-retest) analyses.
Changes in the dynamic visual acuity | Immediately after the vestibular electrodes are activated
  During the experiments, participants have to read aloud sequences of Sloan optotypes of decreasing size displayed in a random order one at a time on a computer screen . The sequence starts with a five letters presentation at 1 logMAR (logarithm of the Minimum Angle of Resolution). If the letter recognition rate is above chance (>10%), the letter size is decreased by a step of 0.1 logMAR and five new letters are presented one at a time. The experiments is carried out on a treadmill either in statoc or in dynamic (fastest walking speed as possible) condition.
Changes in angular error during a navigation task | Immediately after the vestibular electrodes are activated
  Participants will perform a path integration or 'complete the triangle' virtual reality task in which the subject moves in a virtual environment toward two visual targets following each other and then has to come-back to his starting point. The angular error can then be calculated.
Changes in orthostatic hypotension test results (Shellong test) | Before and immediately after the vestibular electrodes are activated
  The subject lies on an examination table and is at rest since at least 10mn. Blood pressure and cardiac frequency are measured in lying position. At time zero the subject stands up and his blood pressure and cardiac frequency are then measured at different time points (1mn, 3mn, 5mn and 10mn after time zero). The test will be systematically performed by trained medical staff. All relevant clinical signs of the participant which could appear during the test will be documented.
Changes in pupil size (pupillometry) | Before and immediately after the vestibular electrodes are activated
  Using an eye tracker (EyeLink) to provide a reliable and objective measurement of pupillary size, symmetry, and reactivity through measurement of the pupil light reflex, the investigators will measure changes in pupil size before and right after the activation of the vestibular implant.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Guinand, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutabla A, Cavuscens S, Ranieri M, Cretallaz C, Kingma H, van de Berg R, Guinand N, Perez Fornos A. Simultaneous activation of multiple vestibular pathways upon electrical stimulation of semicircular canal afferents. J Neurol. 2020 Dec;267(Suppl 1):273-284. doi: 10.1007/s00415-020-10120-1. Epub 2020 Aug 10. PMID 32778921
- [Background] Fornos AP, van de Berg R, Armand S, Cavuscens S, Ranieri M, Cretallaz C, Kingma H, Guyot JP, Guinand N. Cervical myogenic potentials and controlled postural responses elicited by a prototype vestibular implant. J Neurol. 2019 Sep;266(Suppl 1):33-41. doi: 10.1007/s00415-019-09491-x. Epub 2019 Aug 8. PMID 31396689
- [Background] Perez Fornos A, Cavuscens S, Ranieri M, van de Berg R, Stokroos R, Kingma H, Guyot JP, Guinand N. The vestibular implant: A probe in orbit around the human balance system. J Vestib Res. 2017;27(1):51-61. doi: 10.3233/VES-170604. PMID 28387690
- [Background] Cretallaz C, Boutabla A, Cavuscens S, Ranieri M, Nguyen TAK, Kingma H, Van De Berg R, Guinand N, Perez Fornos A. Influence of systematic variations of the stimulation profile on responses evoked with a vestibular implant prototype in humans. J Neural Eng. 2020 Jun 12;17(3):036027. doi: 10.1088/1741-2552/ab8342. PMID 32213673
- [Background] Guinand N, Van de Berg R, Cavuscens S, Stokroos R, Ranieri M, Pelizzone M, Kingma H, Guyot JP, Perez Fornos A. Restoring Visual Acuity in Dynamic Conditions with a Vestibular Implant. Front Neurosci. 2016 Dec 22;10:577. doi: 10.3389/fnins.2016.00577. eCollection 2016. PMID 28066163
- [Background] Guinand N, Van de Berg R, Cavuscens S, Ranieri M, Schneider E, Lucieer F, Kingma H, Guyot JP, Perez Fornos A. The Video Head Impulse Test to Assess the Efficacy of Vestibular Implants in Humans. Front Neurol. 2017 Nov 14;8:600. doi: 10.3389/fneur.2017.00600. eCollection 2017. PMID 29184530
- [Background] van de Berg R, Guinand N, Nguyen TA, Ranieri M, Cavuscens S, Guyot JP, Stokroos R, Kingma H, Perez-Fornos A. The vestibular implant: frequency-dependency of the electrically evoked vestibulo-ocular reflex in humans. Front Syst Neurosci. 2015 Jan 20;8:255. doi: 10.3389/fnsys.2014.00255. eCollection 2014. PMID 25653601
- [Background] Nguyen TAK, Cavuscens S, Ranieri M, Schwarz K, Guinand N, van de Berg R, van den Boogert T, Lucieer F, van Hoof M, Guyot JP, Kingma H, Micera S, Perez Fornos A. Characterization of Cochlear, Vestibular and Cochlear-Vestibular Electrically Evoked Compound Action Potentials in Patients with a Vestibulo-Cochlear Implant. Front Neurosci. 2017 Nov 21;11:645. doi: 10.3389/fnins.2017.00645. eCollection 2017. PMID 29209162
- [Background] Perez Fornos A, Guinand N, van de Berg R, Stokroos R, Micera S, Kingma H, Pelizzone M, Guyot JP. Artificial balance: restoration of the vestibulo-ocular reflex in humans with a prototype vestibular neuroprosthesis. Front Neurol. 2014 Apr 29;5:66. doi: 10.3389/fneur.2014.00066. eCollection 2014. PMID 24808890
- [Background] Guinand N, van de Berg R, Cavuscens S, Stokroos RJ, Ranieri M, Pelizzone M, Kingma H, Guyot JP, Perez-Fornos A. Vestibular Implants: 8 Years of Experience with Electrical Stimulation of the Vestibular Nerve in 11 Patients with Bilateral Vestibular Loss. ORL J Otorhinolaryngol Relat Spec. 2015;77(4):227-240. doi: 10.1159/000433554. Epub 2015 Sep 15. PMID 26367113
- [Background] Pelizzone M, Fornos AP, Guinand N, van de Berg R, Kos I, Stokroos R, Kingma H, Guyot JP. First functional rehabilitation via vestibular implants. Cochlear Implants Int. 2014 May;15 Suppl 1:S62-4. doi: 10.1179/1467010014Z.000000000165. No abstract available. PMID 24869447